CLINICAL TRIAL: NCT03006055
Title: The Detection of Circulating Tumor Cells (CTCs) in Breast Cancer With a Novel in Vivo Device
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Viroad Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIROAD01
Record Dates: First submitted 2016-12-21; First posted 2016-12-30 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Circulating Tumor Cells.Breast

ARMS (2):
- MBC Group (Experimental): metastatic breast cancer Age：18-75 ECOG:0-2
  Interventions: Device: Circulating tumor cells
- Control Group (Experimental): benign breast tumour Age：18-75 ECOG:0-2
  Interventions: Device: Circulating tumor cells

INTERVENTIONS:
Device: Circulating tumor cells

SUMMARY:
The GILUPI CellCollector® is the first in vivo CTC isolation product worldwide which is CE approved. Application data of CellCollector in China is not available now. The purpose of this clinical trial is to confirm the validation and safety of CellCollector in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Metastasis breast cancer confirmed with imaging examination
* Have agreed to undergo CTC analysis in vivo;
* ECOG：0-2

Exclusion Criteria:

* Non-metastasis breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Validation of CellCollector | 6 month
  CTC enumeration and detection rate in Chinese patients with metastasis breast cancer will be analyzed by using CellCollector.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 month
  Number of participants with treatment-related adverse events and blood IgE level will be analyzed after CellCollector application.

CONTACTS AND LOCATIONS:
Locations (1):
- The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality, China